CLINICAL TRIAL: NCT04183179
Title: Happy Family, Healthy Kids: An Intergenerational Program to Promote Healthy Eating Habits
Brief Title: Happy Family, Healthy Kids Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Jiying Ling, Assistant Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Grant #R-1904-144322
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Healthy Diet; Stress; Pediatric Obesity; Intergenerational Relations
Keywords: Obesity prevention; Early childhood; Intergenerational; Healthy eating; Life stress management
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: The program will be evaluated with about 100 Head Start children, aged 3 to 5 years, and their parents (one parent per family) in four urban and three rural Head Start centers to compare the program outcomes between urban and rural settings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Program (Experimental): The 14-week healthy eating program activities including four components:
  1. A 14-week parent Facebook-based program focusing on stress management and healthy eating to reduce emotional eating and increase parents' capacity to initiate healthy eating practices at home
  2. Three parent face-to-face or virtual meetings at Head Start centers to connect parents with each other in person, offer healthy cooking tools/classes, and discuss behavioral change strategies and challenges
  3. 14-week child "Eat My ABCs" program at Head Start centers to provide an age-appropriate, healthy eating program to children
  4. Weekly child letter to parents to connect child learning at the Head Start center with parental practices at home
  Interventions: Behavioral: Happy Family, Healthy Kids Program

INTERVENTIONS:
Behavioral: Happy Family, Healthy Kids Program — The 14-week healthy eating program activities including four components:
  1. A 14-week parent Facebook-based program focusing on stress management and healthy eating to reduce emotional eating and increase parents' capacity to initiate healthy eating practices at home
  2. Three parent face-to-face or virtual meetings at Head Start centers to connect parents with each other in person, offer healthy cooking tools/classes, and discuss behavioral change strategies and challenges
  3. 14-week child "Eat My ABCs" program at Head Start centers to provide an age-appropriate, healthy eating program to children
  4. Weekly child letter to parents to connect child learning at the Head Start center with parental practices at home

SUMMARY:
Happy Family, Healthy Kids program, funded by the Michigan Health Endowment Fund, is a 14-week healthy eating program aimed to foster "Happy Family & Healthy Kids." The program will target parental emotional eating through a life stress management component, and parents will be coached on making happy and healthy eating behavioral changes at home that will support their children to establish lifelong healthy eating habits. At the end of this project, the investigators expect to have an effective, comprehensive, and sustainable healthy eating program ready to expand to any Head Start center in an urban or rural setting.

DETAILED DESCRIPTION:
In Project Year 1, the program will be evaluated with about 100 Head Start children, aged 3 to 5 years, and their parents (one parent per family) in four urban and four rural Head Start centers. The investigators will compare the program outcomes between urban and rural settings. All involved Head Start centers will support MSU staff to conduct data collection activities (e.g., online survey completed by parents; height, weight, and blood pressure measures; hair samples collected from both children and parents). MSU staff, along with Head Start staff, will implement the 14-week healthy eating program activities including four components:

1. A 14-week parent Facebook-based program focusing on stress management and healthy eating to reduce emotional eating and increase parents' capacity to initiate healthy eating practices at home
2. Three parent face-to-face or virtual meetings at Head Start centers to connect parents with each other in person, offer healthy cooking tools/classes, and discuss behavioral change strategies and challenges
3. 14-week child "Eat My ABCs" program at Head Start centers to provide an age-appropriate, healthy eating program to children
4. Weekly child letter to parents to connect child learning at the Head Start center with parental practices at home

In Project Year 2, the investigators will finalize the program based on the evaluation outcomes in Project Year 1, and work closely with the participating Head Start organizations to disseminate the healthy eating program to all the participating Head Start centers and classes.

ELIGIBILITY:
Inclusion Criteria:

There are ten inclusion criteria (five for preschoolers and five for caregivers).

Preschoolers must:

1. Have parental consent.
2. Have child assent if the child is 5 years old.
3. Be 3-5 years of age.
4. Be able to understand and speak English. The intervention will be delivered in English.
5. Be enrolled in the full-day or part-day Head Start program.

Caregivers must:

1. Provide consent.
2. Be the primary adult caregiver (≥ 18 years old) for the preschooler. Primary caregiver refers to the one person most responsible for providing care to the preschooler on a daily basis.
3. Be able to read, understand, and speak English. The intervention will be delivered in English.
4. Have at least weekly Internet access using a smartphone, tablet, or a computer. Each caregiver needs to have Internet access to access the study's Facebook group for participating in the Facebook-based program.
5. Be willing to use Facebook. Since the caregiver intervention component will be delivered via Facebook, caregivers need to be willing to use Facebook in the study.

Exclusion Criteria:

There are three exclusion criteria for both caregivers and preschoolers.

1. Preschoolers or caregivers who have medical conditions precluding participating in dietary changes.
2. Preschoolers or caregivers who have diagnosed health conditions known to impact weight (e.g., Prader-Willi Syndrome) or are taking weight-affecting medications (e.g., stimulants).
3. Preschoolers who have diagnosed developmental disabilities (e.g., autism), or caregivers who have diagnosed psychiatric or mental health problems.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Betsie Valley Elementary, Thompsonville, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data including code book can be shared with other researchers upon request.

REFERENCES:
- [Derived] Ling J, Chen S, Zhang N, Robbins LB, Kerver JM. Happy Family, Healthy Kids: A Healthy Eating and Stress Management Program in Low-Income Parent-Preschooler Dyads. Nurs Res. 2024 Jan-Feb 01;73(1):3-15. doi: 10.1097/NNR.0000000000000697. Epub 2023 Sep 23. PMID 37768980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 107 caregivers and 107 preschoolers were recruited.
Groups:
- Program-Preschoolers: The 14-week healthy eating program activities including 2 components for preschoolers:
  1. 14-week child "Eat My ABCs" program at Head Start centers to provide an age-appropriate, healthy eating program to children
  2. Weekly child letter to parents to connect child learning at the Head Start center with parental practices at home
- Program-Caregivers: The 14-week healthy eating program activities including 2 components for caregivers:
  1. A 14-week parent Facebook-based program focusing on stress management and healthy eating to reduce emotional eating and increase parents' capacity to initiate healthy eating practices at home
  2. Three parent face-to-face or virtual meetings at Head Start centers to connect parents with each other in person, offer healthy cooking tools/classes, and discuss behavioral change strategies and challenges
Period: Overall Study
Arm/Group | Program-Preschoolers | Program-Caregivers
Started (Preschoolers) | 107 | 107 (Caregivers)
Completed | 103 | 103
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: 107 preschoolers and 107 caregivers
Groups:
- Program: The 14-week healthy eating program activities including 4 components:
  1. 14-week child "Eat My ABCs" program at Head Start centers to provide an age-appropriate, healthy eating program to children
  2. Weekly child letter to parents to connect child learning at the Head Start center with parental practices at home
  3. A 14-week parent Facebook-based program focusing on stress management and healthy eating to reduce emotional eating and increase parents' capacity to initiate healthy eating practices at home
  4. Three parent face-to-face or virtual meetings at Head Start centers to connect parents with each other in person, offer healthy cooking tools/classes, and discuss behavioral change strategies and challenges
Arm/Group | Program
Number analyzed (Participants) | 214
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The total sample of 214 include 107 preschoolers and 107 caregivers.
  Years
    Preschoolers: number analyzed (Participants) | 107
    Preschoolers | 3.94 (0.57)
    Caregivers: number analyzed (Participants) | 107
    Caregivers | 30.12 (5.98)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Total 214 participants including 107 preschoolers and 107 caregivers.
  Participants
    Preschoolers: number analyzed (Participants) | 107
    Preschoolers: Female | 58
    Preschoolers: Male | 49
    Caregivers: number analyzed (Participants) | 107
    Caregivers: Female | 102
    Caregivers: Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total 214 participants with 107 preschoolers and 107 caregivers.
  Participants
    Preschooler: number analyzed (Participants) | 107
    Preschooler: Hispanic or Latino | 9
    Preschooler: Not Hispanic or Latino | 98
    Preschooler: Unknown or Not Reported | 0
    Caregivers: number analyzed (Participants) | 107
    Caregivers: Hispanic or Latino | 7
    Caregivers: Not Hispanic or Latino | 100
    Caregivers: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total 214 participants with 107 preschoolers and 107 caregivers.
  Participants
    Preschoolers: number analyzed (Participants) | 107
    Preschoolers: American Indian or Alaska Native | 1
    Preschoolers: Asian | 0
    Preschoolers: Native Hawaiian or Other Pacific Islander | 0
    Preschoolers: Black or African American | 21
    Preschoolers: White | 78
    Preschoolers: More than one race | 7
    Preschoolers: Unknown or Not Reported | 0
    Caregivers: number analyzed (Participants) | 107
    Caregivers: American Indian or Alaska Native | 3
    Caregivers: Asian | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0
    Caregivers: Black or African American | 16
    Caregivers: White | 79
    Caregivers: More than one race | 8
    Caregivers: Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 214

OUTCOME MEASURES:

1. Primary Outcome: Child Dietary Fruit and Vegetable Intake
Description: Child dietary intake will be assessed by the 41-item Block Kids Food Screener. The Block Kids Food Screener is a food frequency questionnaire used to assess dietary intake of fruits, vegetables, dairy, whole grains, protein sources, saturated fat, and added sugars in youth aged 2-17 years old. It has been shown to have significant relationships (r=0.53-0.88) with Nutrition Data System for Research 24-h food recall data. The Block Kids Food Screener has acceptable Cronbach's alphas of 0.76-0.77 for the survey items assessing fruit and vegetable intake among Head Start preschoolers. The completed surveys will be processed and analyzed by NutritionQuest, and the number of cups of fruit and vegetable consumed per day will be used to describe children's fruit and vegetable intake, with a higher number indicating a healthier eating behavior.
Time Frame: Change from baseline child dietary intake at 15 weeks
Population: This outcome is for preschoolers only. Caregivers' outcomes were presented separately.
Measure: Mean (Standard Deviation); unit: Cups per day
Groups:
- Program - Preschooler Participants: The 14-week healthy eating program activities including four components:
  1. A 14-week parent Facebook-based program focusing on stress management and healthy eating to reduce emotional eating and increase parents' capacity to initiate healthy eating practices at home
  2. Three parent face-to-face or virtual meetings at Head Start centers to connect parents with each other in person, offer healthy cooking tools/classes, and discuss behavioral change strategies and challenges
  3. 14-week child "Eat My ABCs" program at Head Start centers to provide an age-appropriate, healthy eating program to children
  4. Weekly child letter to parents to connect child learning at the Head Start center with parental practices at home
  Happy Family, Healthy Kids Program: The 14-week healthy eating program activities including four components:
  1. A 14-week parent Facebook-based program focusing on stress management and healthy eating to reduce emotional eating and increase parents' capacity to initiate healthy eating practices at home
  2. Three parent face-to-face or virtual meetings at Head Start centers to connect parents with each other in person, offer healthy cooking tools/classes, and discuss behavioral change strategies and challenges
  3. 14-week child "Eat My ABCs" program at Head Start centers to provide an age-appropriate, healthy eating program to children
  4. Weekly child letter to parents to connect child learning at the Head Start center with parental practices at home
Arm/Group | Program - Preschooler Participants
Number analyzed (Participants) | 107
Cups per day | 0.07 (1.04)

2. Secondary Outcome: Child Emotional Overeating
Description: Child eating style will be assessed by the 35-item Child Eating Behavior Questionnaire. It has five response choices ranging from 1=never to 5=always. The Child Eating Behavior Questionnaire has eight factors including food responsiveness, emotional overeating, enjoyment of food, desire to drink, satiety responsiveness, slowness in eating, emotional undereating, and food fussiness with good reliability and validity among preschoolers. A mean score (min-max: 1-5) for the emotional overeating factor will be calculated, with a higher mean factor score indicating a higher level of emotional overeating.
Time Frame: Change from baseline to 15 weeks
Measure: Mean (Standard Deviation); unit: Mean score
Arm/Group | Program - Preschooler Participants
Number analyzed (Participants) | 107
Mean score | 0.05 (0.46)

3. Secondary Outcome: Child Body Mass Index Z-score
Description: Height and weight will be measured to the nearest 0.1 cm with a ShorrBoard stadiometer and to the nearest 0.1 kg with a Seca model 874 portable electronic weight scale, respectively. All measurements will occur in a private room with participants removing their shoes, jackets, or heavy clothes. BMI z-score for age and sex will be determined via SAS program for CDC Growth Charts. The BMI Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population. Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population. A negative change in Z-scores indicates a favorable outcome.
Time Frame: Change from baseline body mass index z-score at 15 weeks
Measure: Mean (Standard Deviation); unit: BMI z score
Arm/Group | Program - Preschooler Participants
Number analyzed (Participants) | 107
BMI z score | -0.06 (0.48)

4. Secondary Outcome: Systolic and Diastolic Blood Pressure
Description: Both systolic (SBP) and diastolic blood pressure (DBP) will be measured using the Omron HEM-705-CP digital blood pressure monitor in the right arm of each relaxed (rest at least 15 minutes) and seated participant. The Omron HEM-705-CP can provide accurate estimation of blood pressure in both children and adults with a sensitivity of 82% and specificity of 98%.
Time Frame: Change from baseline blood pressure at 15 weeks
Population: 214 participants include 107 preschoolers and 107 caregivers.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Program: The 14-week healthy eating program activities including four components:
  1. A 14-week parent Facebook-based program focusing on stress management and healthy eating to reduce emotional eating and increase parents' capacity to initiate healthy eating practices at home
  2. Three parent face-to-face or virtual meetings at Head Start centers to connect parents with each other in person, offer healthy cooking tools/classes, and discuss behavioral change strategies and challenges
  3. 14-week child "Eat My ABCs" program at Head Start centers to provide an age-appropriate, healthy eating program to children
  4. Weekly child letter to parents to connect child learning at the Head Start center with parental practices at home
  Happy Family, Healthy Kids Program: The 14-week healthy eating program activities including four components:
  1. A 14-week parent Facebook-based program focusing on stress management and healthy eating to reduce emotional eating and increase parents' capacity to initiate healthy eating practices at home
  2. Three parent face-to-face or virtual meetings at Head Start centers to connect parents with each other in person, offer healthy cooking tools/classes, and discuss behavioral change strategies and challenges
  3. 14-week child "Eat My ABCs" program at Head Start centers to provide an age-appropriate, healthy eating program to children
  4. Weekly child letter to parents to connect child learning at the Head Start center with parental practices at home
Arm/Group | Program
Number analyzed (Participants) | 214
mmHg
  Child SBP: number analyzed (Participants) | 107
  Child SBP | 1.02 (11.77)
  Child DBP: number analyzed (Participants) | 107
  Child DBP | -1.60 (12.38)
  Caregiver SBP: number analyzed (Participants) | 107
  Caregiver SBP | -3.64 (11.96)
  Caregiver DBP: number analyzed (Participants) | 107
  Caregiver DBP | -2.10 (9.21)

5. Other Pre Specified Outcome: Parental Knowledge of Health Eating
Description: Parental knowledge of health eating will be assessed by the 10-item Parental Nutrition Knowledge Scale. This scale has been used with Head Start parents to assess their knowledge level. The sum of the 10 items, with a range from 0 to 10, will be calculated, with a higher sum score indicating greater knowledge on healthy eating and physical activity.
Time Frame: Change from baseline parental knowledge of health eating at 15 weeks
Measure: Mean (Standard Deviation); unit: Sum score on a scale
Arm/Group | Program
Number analyzed (Participants) | 107
Sum score on a scale | 0.44 (1.21)

6. Other Pre Specified Outcome: Parental Self-efficacy for Supporting Health Eating
Description: Parental self-efficacy for supporting health eating will be assessed with the 12-item Parental Eating Self-Efficacy Scale. The scale has shown to have a good internal consistency reliability of 0.94 with Head Start parents. The mean score of the 12 items, with a range from 0 to 10, will be calculated, with a higher mean score indicating greater self-efficacy.
Time Frame: Change from baseline parental self-efficacy for supporting health eating at 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program
Number analyzed (Participants) | 107
score on a scale | 0.56 (1.25)

7. Other Pre Specified Outcome: Parental Support for Health Eating
Description: Parental support for health eating will be measured by the 7-item Parental Support Scale for Eating Habits. A prior study with Head Start parents showed that the scale had a Cronbach's alpha of 0.87. The mean score of the seven items, with a range from 1 to 6, will be calculated, with a higher mean score indicating greater parental support.
Time Frame: Change from baseline parental support for health eating at 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program
Number analyzed (Participants) | 107
score on a scale | 0.47 (0.89)

8. Other Pre Specified Outcome: Parental Feeding Practice Skill
Description: Parental feeding practice skill will be assessed by the Child Feeding Questionnaire. The Child Feeding Questionnaire has seven factors: perceived responsibility, perceived caregiver weight, perceived child weight, concerns about child weight, restriction, pressure to eat, and monitoring with good Cronbach's alphas of 0.73, 0.80, 0.75, 0.73, 0.69, 0.65, and 0.82 among Head Start parents, respectively. The mean score of the items for each factor, with a range from 1 to 5, will be calculated, with a higher mean score indicating greater perceived responsibility, perceived caregiver weight, perceived child weight, concerns about child weight, pressure to eat, restriction, and monitoring, respectively.
Time Frame: Change from baseline parental feeding practice skill at 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program
Number analyzed (Participants) | 107
score on a scale
  perceived responsibility | -0.05 (0.45)
  perceived caregiver weight | 0.003 (0.37)
  perceived child weight | -0.03 (0.30)
  concerns about child weight | 0.02 (0.44)
  restriction | -0.09 (0.79)
  pressure to eat | -0.11 (0.78)
  monitoring | 0.04 (1.07)

9. Other Pre Specified Outcome: Parental Perceived Stress
Description: Parental perceived stress will be assessed by the 10-item Perceived Stress Scale (PSS). Literature has support that the 10-item PSS has better psychometric properties than the original 14-item PSS. It has five response choices from 0=never to 4=very often. The sum score of the 10 items will be calculated, with a higher sum score indicating a higher perceived stress level.
Time Frame: Change from baseline parental perceived stress at 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program
Number analyzed (Participants) | 107
score on a scale | 3.74 (9.16)

10. Other Pre Specified Outcome: Parental Coping Strategies
Description: Parental coping strategies will be assessed by the 28-item Brief COPE. The Brief COPE measures 14 coping strategies including self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion, and self-blame. It has four response choices from "1=not at all" to "4=a lot". A sum score, range from 2 to 8, for each coping strategy will be calculated, with a higher sum score indicating a higher level of that coping strategy used.
Time Frame: Change from baseline parental coping strategies at 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program
Number analyzed (Participants) | 107
score on a scale
  Problem-focused coping | 0.14 (0.61)
  Emotion-focused coping | -0.01 (0.44)
  Avoidant coping | 0.01 (0.39)

11. Other Pre Specified Outcome: Parent Fruit/Vegetable/Fiber Intake
Description: Parent fruit/vegetable/fiber intake will be assessed by the 7-item Block Fruit/Vegetable/Fiber Screener. The screener had significant relationships with the 1995 Block 100-item Food Frequency Questionnaire (r=0.71 for fruit/vegetable intake and 0.62 for fiber intake). It has good Cronbach's alphas of 0.75-0.76 among Head Start parents. The survey has six response choices ranging from 0=less than one per week to 5=2 or more a day. Following the equations provided by the NutritionQuest, the number of fruit and vegetable servings per day will be calculated to describe parents' fruit and vegetable intake.
Time Frame: Change from baseline parent fruit/vegetable/fiber intake at 15 weeks
Measure: Mean (Standard Deviation); unit: servings per day
Arm/Group | Program
Number analyzed (Participants) | 107
servings per day | 0.12 (1.53)

12. Other Pre Specified Outcome: Parental Emotional Eating
Description: Parental emotional eating will be assessed by the Three-Factor Eating Questionnaire (TFEQ-R18). The TFEQ-R18 has three domains: uncontrolled eating, emotional eating, and cognitive restraint, with Cronbach's alpha coefficients of 0.84, 0.92, and 0.70, respectively, among U.S. healthy weight, overweight, and obese adults. Another study with tumor survivors aged 15-39 years old further supports the reliability and factor structure of the scale. It has four response choices ranging from 1="definitely false" to 4="definitely true". The mean score of each domain will be calculated, with a higher mean score indicating a higher level of uncontrolled eating, emotional eating, and cognitive restraint, respectively.
Time Frame: Change from baseline parental emotional eating at 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program
Number analyzed (Participants) | 107
score on a scale | 0.01 (0.67)

13. Other Pre Specified Outcome: Home Eating Environment
Description: Home eating environment will be assessed by the 10-item Family Nutrition Screening Tool, with good construct validity in young children. Evidence has shown that the healthier home eating environment is related to healthier BMI and lower odds of food insecurity. It has four response choices ranging from 1=never/almost never to 4=very often/always. The sum score of the 10 items, with a range from 10 to 40, will be calculated, with a higher sum score indicating a healthier home environment.
Time Frame: Change from baseline home eating environment at 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program
Number analyzed (Participants) | 107
score on a scale | 0.87 (3.65)

14. Other Pre Specified Outcome: Food Security Status
Description: Food security status in the past 12 months will be assessed by the 18-item U.S. Household Food Security Survey Module. It has two subscales: a 10-item Adult Food Security subscale and an 8-item Child Food Security subscale. Raw score, ranging from 0 to 18, will be calculated for the whole scale, adult subscale, and child subscale, respectively, with a higher raw score indicating a higher level of food insecurity. Household will be categorized as 0-2=food secure and 3-18=food insecure.
Time Frame: Change from baseline food security status at 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program
Number analyzed (Participants) | 107
score on a scale | -0.01 (0.87)

15. Other Pre Specified Outcome: Parent Body Mass Index
Description: Body mass index will be calculated based on weight (kg)/height (m2). Data collection procedures for parents will be similar to those employed for preschoolers.
Time Frame: Change from baseline parent proportion of overweight and obesity and body mass index at 15 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Program
Number analyzed (Participants) | 107
kg/m^2 | -0.13 (3.40)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed and collected throughout the entire study during baseline data collection, intervention implementation, and post-intervention data collection lasting for about 1 year and 4 months.
Groups:
- Program for Preschoolers: The 14-week healthy eating program activities including 2 components for preschoolers:
  1. 14-week child "Eat My ABCs" program at Head Start centers to provide an age-appropriate, healthy eating program to children
  2. Weekly child letter to parents to connect child learning at the Head Start center with parental practices at home
- Program for Caregivers: The 14-week healthy eating program activities including 2 components for caregivers:
  1. A 14-week parent Facebook-based program focusing on stress management and healthy eating to reduce emotional eating and increase parents' capacity to initiate healthy eating practices at home
  2. Three parent face-to-face or virtual meetings at Head Start centers to connect parents with each other in person, offer healthy cooking tools/classes, and discuss behavioral change strategies and challenges
Arm/Group | Program for Preschoolers | Program for Caregivers
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/107
Other Adverse Events (participants affected / at risk) | 0/107 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT04183179/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT04183179/SAP_001.pdf